CLINICAL TRIAL: NCT00809601
Title: Randomized Controlled Study of Transmyringeal Tubes
Brief Title: Study of Different Kinds of Ear Tubes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Danderyd Hospital (Other)
Collaborators: Centre for clinical research Vastmanland (Unknown)
Responsible Party: Principal Investigator, Magnus von Unge, Principal investigator, Danderyd Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2008/69-31/3
Record Dates: First submitted 2008-05-02; First posted 2008-12-17 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Recurrent Acute Otitis Media; Otitis Media With Effusion With Hearing Impairment
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Device: Insertion of a specific type of ventilation tube through the tympanic membrane

INTERVENTIONS:
Device: Insertion of a specific type of ventilation tube through the tympanic membrane — The ventilation tubes are tested using one type in one ear and another type as an active comparator in the other ear.
  The investigators will test in total 4 different kinds of tubes. Four different combinations of tubes will be tested.
  The first combination will test:
  "Shepard tube" (double flanged, Fluoroplastic) vs "Donaldson tube" (double flanged, silicone)
  The second combination will test:
  "Straight tube" (single flanged, Fluoroplastic) vs "Armstrong" (single flanged, silicone)
  The third combination will test:
  "Armstrong" (single flanged, silicone) vs "Donaldson tube" (double flanged, silicone)
  The fourth combination will test:
  "Straight tube" (single flanged, Fluoroplastic) vs "Shepard tube" (double flanged, Fluoroplastic)

SUMMARY:
There are different kinds of ear tubes that may be inserted into the tympanic membrane to relieve recurrent acute otitis and hearing impairment due to otitis media with effusion. The tubes differ in size, shape and material.

No-one knows if there are differences between the different kinds of tubes regarding complications.

The investigators' hypothesis is that there is differences between the different kinds of tubes regarding complications.

To test the investigators' hypothesis, the investigators are about to conduct a randomized controlled study of four kinds of tubes having two different material and two different shapes.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1-10 planned for bilateral ventilation tubes

Exclusion Criteria:

* Ongoing ear infection
* Previous insertion of ventilation tube

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2008-05; Primary Completion 2014-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Time to complete expulsion of the ventilation tube from the tympanic membrane | 45 months

SECONDARY OUTCOMES:
Persistent tympanic membrane perforation | 45 months
Need for tube extraction (pain or infection) | 45 months
Pain leading to health care contact | 45 months
Tube related ear infection | 45 months
Obstruction of the tube | 45 months
Presence of myringosclerosis | 45 months

CONTACTS AND LOCATIONS:
Overall Officials: Magnus von Unge, MD, PhD, Principal Investigator — ENT-dept Karolinska Hospital; Johan Knutsson, MD, Study Director — Centre for clinical research Vastmanland
Locations (1):
- Danderyds Hospital, Stockholm, Stockholm County, Sweden